CLINICAL TRIAL: NCT04309734
Title: A Phase I/IIa Study Assessing AT-777 in Healthy Subjects and AT-777 in Combination With AT-527 in HCV-Infected Subjects
Brief Title: Study of AT-777 in Healthy Subjects and AT-777 in Combination With AT-527 in HCV-Infected Subjects
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Withdrawn prior to study initiation.
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: AT-01C-001; 2019-004997-24 (EudraCT Number)
Record Dates: First submitted 2020-03-13; First posted 2020-03-16 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Hepatitis C; Hepatitis C, Chronic; Chronic Hepatitis C; Hepatitis C Virus Infection; HCV Infection
MeSH Terms: conditions — Hepatitis C; Hepatitis C, Chronic | interventions — AT-511

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Part A is randomized, double-blind. Part B is open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A - 60 mg AT-777 single dose (Experimental)
  Interventions: Drug: AT-777
- Part A - 120 mg AT-777 single dose (Experimental)
  Interventions: Drug: AT-777
- Part A - Placebo single dose (Placebo Comparator)
  Interventions: Drug: Placebo
- Part B - 60 mg AT-777 + 550 mg AT-527 once daily for 8 weeks (Experimental)
  Interventions: Drug: AT-777; Drug: AT-527

INTERVENTIONS:
Drug: AT-777 — Administered orally as one or two 60 mg capsule(s) of AT-777 (inhibitor of HCV nonstructural protein 5A (NS5A)), depending on the arm.
  Arms: Part A - 120 mg AT-777 single dose; Part A - 60 mg AT-777 single dose; Part B - 60 mg AT-777 + 550 mg AT-527 once daily for 8 weeks
Drug: Placebo — Administered orally, as one or two placebo capsules, depending on the arm.
  Arms: Part A - Placebo single dose
Drug: AT-527 — Administered orally as one 550 mg tablet of AT-527 (nucleotide prodrug inhibitor of HCV nonstructural protein 5B (NS5B) polymerase), depending on the arm.
  Arms: Part B - 60 mg AT-777 + 550 mg AT-527 once daily for 8 weeks

SUMMARY:
This study has two parts. Part A will assess the safety, tolerability and pharmacokinetics (PK) of AT-777 in healthy subjects. Part B will assess the safety, antiviral activity/efficacy and PK of AT-777 in combination with AT-527 after 8 weeks of treatment in HCV-infected subjects.

ELIGIBILITY:
Inclusion Criteria:

All:

* Body mass index (BMI) of 18-35 kg/m2
* Must agree to use protocol-specified methods of contraception
* Negative pregnancy test
* Willing to comply with the study requirements and to provide written informed consent

Additional for Part A:

-18-55 years of age

Additional for Part B:

* 18-65 years of age
* HCV genotype 1, 2 or 3
* Documented history compatible with chronic hepatitis C
* HCV RNA ≥ 10,000 IU/mL at Screening

Exclusion Criteria:

All:

* Pregnant or breastfeeding
* Abuse of alcohol or drugs
* Use of other investigational drugs within 30 days of dosing
* Other clinically significant medical conditions

Additional for Part B:

* Prior exposure to any HCV NS5A inhibitor
* Cirrhosis
* Co-infection with hepatitis B virus or HIV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Through Day 6 for subjects in Part A
  Number of subjects experiencing treatment-emergent adverse events
Incidence of Treatment-Emergent Adverse Events | Through 4 weeks after end of treatment for subjects in Part B
  Number of subjects experiencing treatment-emergent adverse events
Antiviral Activity of AT-777 and AT-527 | Through 2 weeks of treatment for subjects in Part B
  Number of subjects who achieve plasma HCV RNA < lower limit of quantitation (LLOQ) and target not detected (TND)

SECONDARY OUTCOMES:
AT-777 maximum plasma concentration (Cmax) | Day 1 for subjects in Part A
  PK
AT-777 area under the concentration-time curve (AUC) | Day 1 for subjects in Part A
  PK
Proportion of subjects achieving sustained virologic response (SVR) | 12 weeks after end of treatment for subjects in Part B
  SVR defined as the HCV RNA < lower limit of quantitation (LLOQ) at 12 weeks after end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Jian Zhou, Study Director — Atea Pharmaceuticals
Locations (1):
- Clinical Trial Site, Antwerp, Belgium